CLINICAL TRIAL: NCT07206446
Title: A Prospective Evaluation of a Prescription Digital Therapeutic for Treatment of Overactive Bladder in Women: The RiSolve Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Galway (Other)
Collaborators: Enterprise Ireland (Other Government)
Responsible Party: Principal Investigator, Andrew Murphy, Foundation Professor, University of Galway
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNI-2023-007; CIV-25-08-054117 (Other: Health Products Regulatory Authority (EUDAMED ID))
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Overactive Bladder (OAB); Over Active Bladder
Keywords: Over active bladder; urogynaecology; prescription digital therapeutic; pdtx; app; mobile app; decentralized; decentralised
MeSH Terms: conditions — Urinary Bladder, Overactive; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental): All participants meeting criteria for inclusion and not exclusion will be given access to the app
  Interventions: Device: RiSolve

INTERVENTIONS:
Device: RiSolve — RiSolve is a Class I device in accordance with Rule 11 of Annex VIII of EU Medical Device Regulation (MDR) 2017/745. The RiSolve App is a smartphone application that users can download following a diagnosis of OAB by a healthcare provider, and following prescription of the RiSolve App. RiSolve consists of an 8-week program including activities to set baselines and assess progress, treatment modules, and modules to enhance engagement.
  As part of setting baselines and assessing progress, participants complete a series of clinically validated questionnaires. This data is presented to users to promote self-monitoring of behaviours and a deeper understanding of their symptoms. A patient report is auto-generated at the end of treatment. This is sent to the patient and contains their in-app self-generated data, their questionnaire results and their bladder diary data (see Appendix 1: RiSolve Patient Report). This information is also provided to the prescribing healthcare provider as an object

SUMMARY:
The RiSolve Trial is a prospective, single-arm, post-market clinical investigation designed to evaluate the effectiveness, usability, and safety of a prescription digital therapeutic (PDTx) for women suffering from overactive bladder (OAB). The study is sponsored by the University of Galway and led by Professor Andrew W. Murphy. It is scheduled to begin in August 2025 and conclude in March 2026, and will be conducted through the Primary Care Clinical Trials Network at the University of Galway. Sixty adult women based in the Republic of Ireland will be recruited to take part. Eligible participants must be at least eighteen years old, fluent in English, own a smartphone, and report bothersome OAB or urgency incontinence symptoms. Women who are pregnant, receiving certain bladder-related treatments, or using specific medications or devices will be excluded.

Overactive bladder is a chronic condition defined by urgency, urinary frequency, nocturia, and often urgency incontinence. It is highly prevalent among women and significantly impacts quality of life, with effects ranging from sleep disruption to reduced occupational performance and heightened risks of anxiety and depression. Standard treatment guidelines recommend a tiered approach, beginning with behavioural therapy, followed by pharmacological options, and finally invasive procedures such as Botox injections or neuromodulation. Behavioural therapy, although considered the gold standard, is often difficult for patients to access due to limited provider availability, cost, and stigma. RiSolve was developed to overcome these barriers by offering a comprehensive, digital, prescription-only therapeutic program.

The investigational device, the RiSolve App (REF: PDTxA001), is a CE-marked Class I medical device developed in accordance with the EU Medical Device Regulation (MDR 2017/745). It delivers an eight-week structured program combining behavioural therapy with a novel digital cognitive behavioural therapy component. Content includes bladder training, pelvic floor exercises, urge suppression strategies, education on bladder health and diet, and general wellbeing modules covering sleep, stress, and exercise. The app also provides interactive tools such as quizzes, bladder diaries, and personalised feedback. Patients complete clinically validated questionnaires and receive auto-generated progress reports, which are also shared with healthcare providers. In its design, RiSolve builds on earlier pilot work with a prior app developed at the University of Galway, which demonstrated improvements in OAB symptoms and quality of life.

The primary aim of the study is to assess usability of the RiSolve App, measured using the user version of the Mobile Application Rating Scale (uMARS). Secondary objectives include evaluating symptom improvement using the Overactive Bladder Questionnaire short-form Symptom Severity scale (OAB-q SF SS) and assessing quality of life changes with the OAB-q SF HQoL scale. Safety outcomes will focus on identifying any device-related serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult women aged 18 and older with bothersome OAB symptoms: (i.e. must answer YES to one of the following):

  * Do you have a sudden need to rush to the toilet to urinate that is bothersome? OR
  * Does urine leak before you can get to the toilet?
* Fluency and literacy in English to enable them to understand and complete treatment and required assessments
* Currently based in the Republic of Ireland
* Ownership and use of a smartphone
* Use of at least one mobile App
* Willing to forego commencing any other OAB treatments outside of RiSolve for the trial treatment period.

Exclusion Criteria:

* Current use of an anticholinergic/beta-agonist, within the previous two weeks and/or at the date of consenting

  * Currently using intermittent or indwelling catheter
  * Currently pregnant or planning pregnancy during the study treatment period
  * Currently receiving treatment for bladder/urethral, colon/anal, or cervical cancer
  * Voiding dysfunction (i.e. if Yes is an answer to any of the following):

    * Do you have pain in your bladder? OR
    * Do you have to strain to urinate?
  * Currently using sacral or tibial neuromodulation.
  * Has had intradetrusor therapy
  * Currently taking antibiotics/drugs for urinary tract infection
  * Planning surgery for pelvic organ prolapse within the trial treatment period
  * Planning to undergo pessary fitting during the study period (Note: patients with an existing pessary are eligible) within the trial treatment period
  * Visual impairment such that in the opinion of the PI would impair their use of the app

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Protocol specifies women
Enrollment: 45 (Estimated)
Dates: Start 2025-09-29 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Usability | From enrollment to the end of treatment at 8-10 weeks
  Usability as measured by the User version of the Mobile Application Rating Scale (uMARS)

SECONDARY OUTCOMES:
Improvement in symptoms | From enrollment to the end of treatment at 8-10 weeks
  Improvement in symptoms, as measured on the Overactive Bladder Questionnaire-Short Form, Symptom Severity (OABq-SF SS) scale
Improvement in quality of life | From enrollment to the end of treatment at 8-10 weeks
  Improvement in quality of life, as measured by the Overactive Bladder Questionnaire-Short Form, health-related quality of life scale (OABq-SF HQoL)

OTHER OUTCOMES:
Device related serious adverse events | From enrollment to the end of treatment at 8-10 weeks
  Number of device related serious adverse events

IPD SHARING:
Plan to Share IPD: No
Proprietary data, sharing would give up competitive advantage

REFERENCES:
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Wilson H. Development and Validation of the User Version of the Mobile Application Rating Scale (uMARS). JMIR Mhealth Uhealth. 2016 Jun 10;4(2):e72. doi: 10.2196/mhealth.5849. PMID 27287964
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Malmstrom TK, Morley JE. SARC-F: a simple questionnaire to rapidly diagnose sarcopenia. J Am Med Dir Assoc. 2013 Aug;14(8):531-2. doi: 10.1016/j.jamda.2013.05.018. Epub 2013 Jun 25. No abstract available. PMID 23810110
- [Background] Dennerstein L, Lehert P, Dudley E. Short scale to measure female sexuality: adapted from McCoy Female Sexuality Questionnaire. J Sex Marital Ther. 2001 Jul-Sep;27(4):339-51. doi: 10.1080/009262301317081098. PMID 11441518
- [Background] Coyne KS, Matza LS, Thompson CL, Kopp ZS, Khullar V. Determining the importance of change in the overactive bladder questionnaire. J Urol. 2006 Aug;176(2):627-32; discussion 632. doi: 10.1016/j.juro.2006.03.088. PMID 16813906
- [Background] Coyne KS, Matza LS, Thompson CL. The responsiveness of the Overactive Bladder Questionnaire (OAB-q). Qual Life Res. 2005 Apr;14(3):849-55. doi: 10.1007/s11136-004-0706-1. PMID 16022077
- [Background] Coyne KS, Thompson CL, Lai JS, Sexton CC. An overactive bladder symptom and health-related quality of life short-form: validation of the OAB-q SF. Neurourol Urodyn. 2015 Mar;34(3):255-63. doi: 10.1002/nau.22559. Epub 2014 Jan 13. PMID 25783168
- [Background] Brookes ST, Donovan JL, Wright M, Jackson S, Abrams P. A scored form of the Bristol Female Lower Urinary Tract Symptoms questionnaire: data from a randomized controlled trial of surgery for women with stress incontinence. Am J Obstet Gynecol. 2004 Jul;191(1):73-82. doi: 10.1016/j.ajog.2003.12.027. PMID 15295345
- [Background] Sanderson DJ, Zavez A, Meekins AR, Eddib A, Lee TG, Barber MD, Duecy E. The Patient Acceptable Symptom State in Female Urinary Incontinence. Female Pelvic Med Reconstr Surg. 2022 Jan 1;28(1):33-39. doi: 10.1097/SPV.0000000000001055. PMID 34009829
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Bradley CS, Rovner ES, Morgan MA, Berlin M, Novi JM, Shea JA, Arya LA. A new questionnaire for urinary incontinence diagnosis in women: development and testing. Am J Obstet Gynecol. 2005 Jan;192(1):66-73. doi: 10.1016/j.ajog.2004.07.037. PMID 15672005
- [Background] Sooknarine C, Farrell S, Sarma S, Salameh F, Burke N, Staunton B, Carr E, Sexton K, Agnew G, Downey A, D'Arcy F, Cundiff GW. Pilot Study of a Digital Behavioral Therapy for Overactive Bladder in Women. Urogynecology (Phila). 2024 Dec 1;30(12):956-961. doi: 10.1097/SPV.0000000000001499. Epub 2024 May 7. PMID 38465995
- [Background] Price JR, Mitchell E, Tidy E, Hunot V. Cognitive behaviour therapy for chronic fatigue syndrome in adults. Cochrane Database Syst Rev. 2008 Jul 16;2008(3):CD001027. doi: 10.1002/14651858.CD001027.pub2. PMID 18646067
- [Background] Etzelmueller A, Vis C, Karyotaki E, Baumeister H, Titov N, Berking M, Cuijpers P, Riper H, Ebert DD. Effects of Internet-Based Cognitive Behavioral Therapy in Routine Care for Adults in Treatment for Depression and Anxiety: Systematic Review and Meta-Analysis. J Med Internet Res. 2020 Aug 31;22(8):e18100. doi: 10.2196/18100. PMID 32865497
- [Background] Melotti IGR, Juliato CRT, Coelho SCA, Lima M, Riccetto CLZ. Is There Any Difference Between Depression and Anxiety in Overactive Bladder According to Sex? A Systematic Review and Meta-Analysis. Int Neurourol J. 2017 Sep;21(3):204-211. doi: 10.5213/inj.1734890.445. Epub 2017 Sep 12. PMID 28954462
- [Background] Harvey J, Finney S, Stewart L, Gillespie J. The relationship between cognition and sensation in determining when and where to void: the concept of cognitive voiding. BJU Int. 2012 Dec;110(11):1756-61. doi: 10.1111/j.1464-410X.2012.11078.x. Epub 2012 May 29. PMID 22642959
- [Background] Olivera CK, Meriwether K, El-Nashar S, Grimes CL, Chen CC, Orejuela F, Antosh D, Gleason J, Kim-Fine S, Wheeler T, McFadden B, Balk EM, Murphy M; Systematic Review Group for the Society of Gynecological Surgeons. Nonantimuscarinic treatment for overactive bladder: a systematic review. Am J Obstet Gynecol. 2016 Jul;215(1):34-57. doi: 10.1016/j.ajog.2016.01.156. Epub 2016 Feb 4. PMID 26851599
- [Background] Norton JM, Dodson JL, Newman DK, Rogers RG, Fairman AD, Coons HL, Star RA, Bavendam TG. Nonbiologic factors that impact management in women with urinary incontinence: review of the literature and findings from a National Institute of Diabetes and Digestive and Kidney Diseases workshop. Int Urogynecol J. 2017 Sep;28(9):1295-1307. doi: 10.1007/s00192-017-3400-x. Epub 2017 Jul 3. PMID 28674734
- [Background] La Rosa VL, Duarte de Campos da Silva T, Rosa de Oliveira A, Marques Cerentini T, Viana da Rosa P, Telles da Rosa LH. Behavioral therapy versus drug therapy in individuals with idiopathic overactive bladder: A systematic review and meta-analysis. J Health Psychol. 2020 Apr;25(5):573-585. doi: 10.1177/1359105319891629. Epub 2019 Dec 3. PMID 31793816
- [Background] Funada S, Watanabe N, Goto T, Negoro H, Akamatsu S, Uozumi R, Kishimoto S, Ichioka K, Segawa T, Furukawa TA, Ogawa O. Clinical feasibility and acceptability of adding cognitive behavioral therapy to pharmacotherapy for drug-resistant overactive bladder in women: A single-arm pilot study. Low Urin Tract Symptoms. 2021 Jan;13(1):69-78. doi: 10.1111/luts.12333. Epub 2020 Jul 3. PMID 32618414
- [Background] Tse V, King J, Dowling C, English S, Gray K, Millard R, O'Connell H, Pillay S, Thavaseelan J; Urological Society of Australia and New Zealand; Urogynaecological Society of Australasia. Conjoint Urological Society of Australia and New Zealand (USANZ) and Urogynaecological Society of Australasia (UGSA) Guidelines on the management of adult non-neurogenic overactive bladder. BJU Int. 2016 Jan;117(1):34-47. doi: 10.1111/bju.13246. Epub 2015 Oct 12. PMID 26456313
- [Background] Corcos J, Przydacz M, Campeau L, Gray G, Hickling D, Honeine C, Radomski SB, Stothers L, Wagg A, Lond F. CUA guideline on adult overactive bladder. Can Urol Assoc J. 2017 May;11(5):E142-E173. doi: 10.5489/cuaj.4586. Epub 2017 May 9. No abstract available. PMID 28503229
- [Background] Nambiar AK, Arlandis S, Bo K, Cobussen-Boekhorst H, Costantini E, de Heide M, Farag F, Groen J, Karavitakis M, Lapitan MC, Manso M, Arteaga SM, Riogh ANA, O'Connor E, Omar MI, Peyronnet B, Phe V, Sakalis VI, Sihra N, Tzelves L, van Poelgeest-Pomfret ML, van den Bos TWL, van der Vaart H, Harding CK. European Association of Urology Guidelines on the Diagnosis and Management of Female Non-neurogenic Lower Urinary Tract Symptoms. Part 1: Diagnostics, Overactive Bladder, Stress Urinary Incontinence, and Mixed Urinary Incontinence. Eur Urol. 2022 Jul;82(1):49-59. doi: 10.1016/j.eururo.2022.01.045. Epub 2022 Feb 23. PMID 35216856
- [Background] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Background] Wu EQ, Birnbaum H, Marynchenko M, Mareva M, Williamson T, Mallett D. Employees with overactive bladder: work loss burden. J Occup Environ Med. 2005 May;47(5):439-46. doi: 10.1097/01.jom.0000161744.21780.c1. PMID 15891521
- [Background] Coyne KS, Sexton CC, Thompson CL, Clemens JQ, Chen CI, Bavendam T, Dmochowski R. Impact of overactive bladder on work productivity. Urology. 2012 Jul;80(1):97-103. doi: 10.1016/j.urology.2012.03.039. PMID 22748868
- [Background] Coyne KS, Sexton CC, Clemens JQ, Thompson CL, Chen CI, Bavendam T, Dmochowski R. The impact of OAB on physical activity in the United States: results from OAB-POLL. Urology. 2013 Oct;82(4):799-806. doi: 10.1016/j.urology.2013.05.035. Epub 2013 Aug 14. PMID 23953610
- [Background] Yehoshua A, Chancellor M, Vasavada S, Malone DC, Armstrong EP, Joshi M, Campbell K, Pulicharam R. Health Resource Utilization and Cost for Patients with Incontinent Overactive Bladder Treated with Anticholinergics. J Manag Care Spec Pharm. 2016 Apr;22(4):406-13. doi: 10.18553/jmcp.2016.22.4.406. PMID 27023694
- [Background] Vrijens D, Drossaerts J, van Koeveringe G, Van Kerrebroeck P, van Os J, Leue C. Affective symptoms and the overactive bladder - a systematic review. J Psychosom Res. 2015 Feb;78(2):95-108. doi: 10.1016/j.jpsychores.2014.11.019. Epub 2014 Nov 27. PMID 25499886
- [Background] Kinsey D, Pretorius S, Glover L, Alexander T. The psychological impact of overactive bladder: A systematic review. J Health Psychol. 2016 Jan;21(1):69-81. doi: 10.1177/1359105314522084. Epub 2014 Mar 2. PMID 24591118
- [Background] Stewart WF, Minassian VA, Hirsch AG, Kolodner K, Fitzgerald M, Burgio K, Cundiff GW, Blaivas J, Newman D, Lerch VR, Dilley A. Predictors of variability in urinary incontinence and overactive bladder symptoms. Neurourol Urodyn. 2010 Mar;29(3):328-35. doi: 10.1002/nau.20753. PMID 19693956
- [Background] Wadensten T, Nystrom E, Nord A, Lindam A, Sjostrom M, Samuelsson E. App-based self-management of urgency and mixed urinary incontinence in women: One-year follow-up. Neurourol Urodyn. 2022 Apr;41(4):945-954. doi: 10.1002/nau.24898. Epub 2022 Mar 9. PMID 35266189
- [Background] Shamliyan T, Wyman J, Bliss DZ, Kane RL, Wilt TJ. Prevention of urinary and fecal incontinence in adults. Evid Rep Technol Assess (Full Rep). 2007 Dec;(161):1-379. PMID 18457475
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- See also: Study webpage featuring downloadable Participant Information Leaflet — https://primarycaretrials.ie/risolve/